CLINICAL TRIAL: NCT04673604
Title: Changing From Preserved, to Preservative-free Cyclosporine 0.1% Enhanced Triple Glaucoma Therapy: Impact on the Rate and Severity of Ocular Surface Disease
Brief Title: From Preserved, to Preservative-free Cyclosporine 0.1% Enhanced Triple Glaucoma Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, AGP Konstas, Professor in Ophthalmology, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 399
Record Dates: First submitted 2020-12-11; First posted 2020-12-17 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Glaucoma; Ocular Surface Disease
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Intervention Model Description: Masked, prospective, placebo-controlled, crossover trial of glaucoma patients with moderate to severe GTR-OSD on preserved latanoprost and dorzolamide/timolol fixed combination therapy for well-controlled open-angle glaucoma was conducted. Patients were randomized to receive preservative-free tafluprost and dorzolamide/timolol fixed combination with either topical placebo or cyclosporine 0.1% for 6 months and will then be crossed over to the opposite therapy. Oxford score of staining will be the primary outcome; osmolarity, matrix-metalloproteinase-9 testing (MMP-9), meibomian gland dysfunction (MGD), adverse events and diurnal intraocular pressure (IOP) comprise the secondary outcomes.
Who Masked: Outcomes Assessor
Masking Description: Only the dosing coordinator is aware of the treatment patients use.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Triple preservative-free therapy with placebo in the evening (Placebo Comparator): In this arm subjects will be randomized to topical therapy comprising preservative-free tafluprost drops dosed in the evening (20:30) and dorzolamide/timolol fixed combination drops administered twice daily (8:00 and 20:00). Patients will use placebo (artificial tears) in the evening (21:00) for 6 months. At the end of this period patients will be crossed over to the other therapy (cyclosporine 0.1% in the evening)
  Interventions: Diagnostic Test: Assessment of ocular surface staining (Oxford score 0-15 scale); Drug: mean diurnal intraocular pressure-lowering
- Triple preservative-free therapy with cyclosporine 0.1% in the evening (Active Comparator): In this arm subjects will be randomized to topical therapy comprising preservative-free tafluprost drops dosed in the evening (20:30) and dorzolamide/timolol fixed combination drops administered twice daily (8:00 and 20:00). Patients will use cyclosporine 0.1% drops in the evening (21:00) for 6 months. At the end of this period all patients will be crossed over to the other therapy (placebo in the evening)
  Interventions: Diagnostic Test: Assessment of ocular surface staining (Oxford score 0-15 scale); Drug: mean diurnal intraocular pressure-lowering

INTERVENTIONS:
Diagnostic Test: Assessment of ocular surface staining (Oxford score 0-15 scale) — Corneal and conjunctiva staining will be recorded according to the Oxford grading scheme for ocular staining (0-15 score).
Drug: mean diurnal intraocular pressure-lowering — At the end of each 6-month period patients will undergo diurnal intraocular pressure assessment with both therapies.

SUMMARY:
There is a lack of evidence on the impact of switching from a combined preserved anti-glaucoma regimen to a preservative-free (PF) one, while employing sufficiently robust OSD metrics. The investigators have therefore carried out a single center, prospective, crossover investigation to compare the 6-month effect of switching well controlled open-angle glaucoma patients with at least moderate glaucoma therapy-related ocular surface disease from preserved to triple preservative-free therapy with and without cyclosporine 0.1% dosed in the evening.

DETAILED DESCRIPTION:
Halting and reversing glaucoma therapy-related ocular surface disease (GTR-OSD) will improve the success of long-term medical therapy, impacting millions of patients worldwide. Chronic medical therapy for glaucoma may be immensely benefitted by limiting disabling GTR-OSD, which would aid in the prevention of blindness. In 2015 a novel cationic formulation of cyclosporine A 0.1% was approved with once in the evening dosing in Europe. It is an effective, targeted immunomodulatory compound reducing inflammatory mediators and providing healing of the ocular epithelium. There remains however a paucity of published controlled evidence for GTR-OSD patients treated with this formulation. In addition, there is a lack of evidence on the impact of switching from a combined preserved anti-glaucoma regimen, to a preservative-free one, while employing sufficiently robust OSD metrics. The investigators have therefore carried out a single center prospective, crossover investigation to compare the 6-month effect of switching well controlled open-angle glaucoma patients with at least moderate GTR-OSD, from preserved to triple PF therapy with and without PF cyclosporine 0.1% dosed in the evening.

ELIGIBILITY:
Inclusion criteria

* Adult patients with well controlled open-angle glaucoma
* Patients chronically treated for more than 6 months with preserved, branded, or generic, triple antiglaucoma therapy comprising latanoprost and dorzolamide/timolol fixed combination
* Subjects should have experienced at least 1 symptom of dry eye (soreness, scratchiness, dryness, grittiness, and burning)
* Additionally, patients should demonstrate at least one of the objective signs for OSD at baseline: positive conjunctival staining with lissamine green and/or evidence of positive corneal staining with fluorescein (assessed with the 15-point Oxford scale),
* Patients must show a BUT<8 seconds
* On screening patients should show a Schirmer test without anesthesia (Schirmer-I test) ≥3 and ≤10 mm in 5 minutes.
* When both eyes qualify the worse eye will be included in the study.

Exclusion criteria

* Best corrected visual acuity <1/10
* Patients with severe dry eye disease or Sjogren's disease
* Presence of eyelid abnormality, corneal disorder or abnormality, ocular surface metaplasia, filamentous keratitis, or corneal neovascularization
* Patients who have undergone ocular surgery (of any type, including laser surgery), or ocular trauma within 4 months prior to screening
* Subjects who had punctal occlusion, or diathermy within 3 months prior to screening or abnormality of the nasolacrimal drainage apparatus.
* Known allergy, or sensitivity to any of the study medications
* Uncontrolled systemic disease, or history or active signs of ocular trauma, infection, inflammation, allergic disease, or herpes; corneal ulcers; recurrent erosions; or uveitis
* Female patients will be excluded if they are pregnant, breastfeeding, planning a pregnancy, or are unwilling to use a reliable form of contraception.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-05-06 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-06-29 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in ocular staining (Oxford score) | 6 months
  The primary efficacy endpoint for this crossover study will be the mean change from baseline in the total ocular staining score as determined by the 15-point Oxford scale of staining on the study eye.

SECONDARY OUTCOMES:
Mean diurnal IOP | 6 months
  Mean diurnal intraocular pressure with the two preservative-free therapies versus preserved baseline will be evaluated as secondary endpoint.
Osmolarity | 6-months
  Mean tear osmolarity with the two PF therapies versus preserved baseline will be evaluated as secondary endpoint.
Matrix-metalloproteinase-9 (MMP-9) over-expression | 6 months
  Mean MMP-9 over-expression with the two PF therapies versus preserved baseline will be evaluated as secondary endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Katsanos, MD, PhD, Study Director — University of Ioannina
Locations (1):
- University Department of Ophthalmology, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No